CLINICAL TRIAL: NCT02240823
Title: Phase 1 Study. Can Fat Derived Stem Cells (SVF) be Used in the Treatment of Erectile Dysfunction After Prostatectomy
Brief Title: Can Fat Derived Stem Cells (SVF) be Used in the Treatment of Erectile Dysfunction After Prostatectomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Martha Haahr M.D (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Martha Haahr M.D, Medical doctor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-Afd-L
Record Dates: First submitted 2014-06-03; First posted 2014-09-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Delayed Graft Function
Keywords: Erectile Function; Mesenchymal Stromal Cells; Stem Cell
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adipose derived stem cells (Experimental)
  Interventions: Other: adipose derived stem cells

INTERVENTIONS:
Other: adipose derived stem cells

SUMMARY:
Prostate cancer is the most common cancer among Danish men, and the incidence is increasing. Studies have shown a high number needed to treat for each saved prostate cancer related death. Since the treatments incur many complications, there is a need to address these. After prostatectomy, 80% experience erectile dysfunction. Sexual life is a central part of people's identity, self-esteem and quality of life. Stem cells have generated a large amount of promising data suggesting that stem cells can alleviate erectile dysfunction, by regenerating nerves as well as endothelial and smooth muscle cells in the corpus cavernous.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer among Danish men, and the incidence is increasing. Studies have shown a high number needed to treat for each saved prostate cancer related death.

After prostatectomy, 80% experience erectile dysfunction. Sexual life is a central part of people's identity, self-esteem and quality of life. Stem cells have generated a large amount of promising data suggesting that stem cells can alleviate erectile dysfunction, by regenerating nerves as well as endothelial and smooth muscle cells in the corpus cavernous.

Animal studies have used stem cell therapy to improve erectile dysfunction in rats after cavernous nerve damage, with invariable high success rate.

In this pilot study will include 30 patient's with erectile dysfunction 3-9 mdr after prostatectomy. The men have no spontaneous erectile function and no response to drug treatment.

Liposuction is carried out in general anesthesia. Isolation of stem cells will be done simultaneously and the stem cells injected into the corpus cavernous directly after the isolation is carried out.

This is a clinical study evaluating an innovative cell therapy procedure.The objective of this study was to evaluate the effects of injection of stem cell of adipose origin.

The project will run over a period of twelve months. Patients will be followed for a period of six months. Treatment efficacy will be assessed from validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Men who have had prostate removed due to prostate cancer regardless bilateral nerve-sparing, unilateral nerve-sparing or non-nerve-sparing surgical technique.
* Erectile dysfunction
* Sexually active/ have sexual interest
* We make no distinction for the patients are operated with

Exclusion Criteria:

* Absence of sexual interest.
* Patients with impaired health condition where anesthesia would be a risk of complications.
* BMI below 20.
* Small amount of abdominal fat assessed by. Ct abdomen.
* Patients on anticoagulant treatment.
* Men with suspicion of residual tumor.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 1 month after surgery
  Adverse Events

SECONDARY OUTCOMES:
Improvement in erectile function, measured i IIEF-5 score | 1,3,6,9 and 12 months
  Assessed by interview and questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Odense Universitet Hospital, Odense, Denmark

REFERENCES:
- [Derived] Haahr MK, Jensen CH, Toyserkani NM, Andersen DC, Damkier P, Sorensen JA, Lund L, Sheikh SP. Safety and Potential Effect of a Single Intracavernous Injection of Autologous Adipose-Derived Regenerative Cells in Patients with Erectile Dysfunction Following Radical Prostatectomy: An Open-Label Phase I Clinical Trial. EBioMedicine. 2016 Jan 19;5:204-10. doi: 10.1016/j.ebiom.2016.01.024. eCollection 2016 Mar. PMID 27077129
- [Derived] Khera M, Albersen M, Mulhall JP. Mesenchymal stem cell therapy for the treatment of erectile dysfunction. J Sex Med. 2015 May;12(5):1105-6. doi: 10.1111/jsm.12871. No abstract available. PMID 25974235